CLINICAL TRIAL: NCT06466811
Title: Identification of Patients at Risk of Undesired Obstruction in External Ventricular Drain: Development of a Score Based on the Extent of Intra-ventricular Hemorrhage. A Single-Center, Prospective Observational Study.
Brief Title: Prediction of Undesired Obstruction in External Ventricular Drains.
Acronym: EVD-OBS
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC24_0074
Record Dates: First submitted 2024-05-14; First posted 2024-06-20 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Intensive Care Unit; Intraventricular Hemorrhage; External Ventricular Drain
Keywords: Intensive care unit; External ventricular drain; Neuromeningeal infection; Obstruction; Intraventricular hemorrhage; Functional outcome
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients of intensive care unit — Patients of intensive care unit having an EVD
Other: Patients of surgical intensive care unit — Patients of surgical intensive care unit having an EVD.

SUMMARY:
Acute obstructive hydrocephalus often complicates intraventricular hemorrhage (IVH). The insertion of an external ventricular drain (EVD) is typically necessary in order to alleviate intracranial pressure by draining excess fluid. However, dysfunction of the EVD whether due to malposition or obstruction, can exacerbate hydrocephalus in an already compromised brain. EVD dysfunction must therefore be promptly detected and treated.

Consequently, identifying high-risk patients and closely monitoring them is imperative. While IVH is known to increase the risk of obstruction in the natural cerebrospinal fluid outflow tract, its association with ventricular drain obstruction remains unproven.

ELIGIBILITY:
Inclusion Criteria :

Patient older than 18 years old,

* admitted to the ICU,
* with first EVD inserted for less than 12 hours,
* and brain imaging (CT or MRI) available in the timespan "24 hours before to 24 hours after" the EVD insertion.

Exclusion Criteria :

* EVD intentionally occluded immediately after its insertion,
* purulent cerebrospinal fluid
* Pregnant or breast-feeding patient
* Moribund patient or patient with decision of withholding or withdrawing life-sustaining treatment within the 12 hours
* Patient with no health insurance
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in an intensive care unit and having an EVD.
Sampling Method: Non-Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the predictive value of IVH severity for EVD obstruction | From EVD insertion to removal up to 100 days.
  HIV severity will be estimated using an adaptation of the existing Graeb's score: the Graeb-EVD score. EVD obstruction is defined by an abnormally reduced drainage flow, requiring intervention to restore normal function (cases of EVD malposition will be excluded).The predictive performance of the Graeb-EVD score will be evaluated by the area under the receiver operating characteristic curve (AUC-ROC). The AUC-ROC ranges from 0 to 1. The predictive ability will be considered acceptable if associated with an AUC-ROC greater than 0.70, good if greater than 0.80, and excellent if greater than 0.90.

SECONDARY OUTCOMES:
To evaluate if HIV is an independent risk factor for the occurrence of at least one episode of unplanned EVD obstruction. | From EVD insertion to removal up to 100 days.
  The researcher will study the risk factors for the occurrence of at least one episode of unplanned EVD obstruction (dependent variable in a logistic regression model) by forcing the inclusion of HIV into this model as an explanatory variable. If the 95% confidence interval of the adjusted odds ratio associated with HIV is greater than 1, HIV will be considered an independent risk factor for unplanned EVD obstruction.
Comparison of the performance of the Graeb-EVD score with that of the original Graeb score and the modified Graeb scores for the prediction of the occurrence of at least one episode of EVD obstruction. | From EVD insertion to removal up to 100 days.
  A p-value of <0.05 in the pairwise comparison of areas under the receiver operating characteristics curves will be used to assert the superiority of the performance of one score over another.
Performance of IVH severity as a predictor of the occurrence of at least one episode of EVD obstruction within the first seven days | From EVD insertion to day 7.
  HIV severity will be estimated using an adaptation of the existing Graeb's score: the Graeb-EVD score. EVD obstruction is defined by an abnormally reduced drainage flow, requiring intervention to restore normal function (cases of EVD malposition will be excluded). The predictive performance of the Graeb-EVD score will be evaluated by the area under the receiver operating characteristic curve (AUC-ROC). The AUC-ROC ranges from 0 to 1. The predictive ability will be considered acceptable if associated with an AUC-ROC greater than 0.70, good if greater than 0.80, and excellent if greater than 0.90.
Evaluation of the 3 Graeb scores (original, modified and EVD) as predictors of the need for a new EVD insertion because of obstruction. | From EVD insertion to hospital discharge up to 12 months.
  The predictive performance of the tested scores will be evaluated by the AUC-ROC. The predictive capacity will be considered acceptable if associated with an AUC-ROC greater than 0.70, good if greater than 0.80, and excellent if greater than 0.90.
Evaluation of the 3 Graeb scores (original, modified and EVD) as predictors of the need for cerebrospinal fluid internal shunt. | From EVD insertion to hospital discharge up to 12 months.
  The predictive performance of the tested scores will be evaluated by the AUC-ROC. The predictive capacity will be considered acceptable if associated with an AUC-ROC greater than 0.70, good if greater than 0.80, and excellent if greater than 0.90.
To evaluate whether the Graeb-EVD, original Graeb, and modified Graeb scores are useful in predicting an unfavorable functional outcome on the day of hospital discharge and at 3±1 months. | From EVD insertion to hospital discharge up to 12 months
  Functional outcome will be considered unfavorable if the modified Rankin scale (ranging from 0 to 6) is 2 or higher, and favorable otherwise. The predictive performance of the tested scores will be evaluated by the AUC-ROC. A score will be considered useful if it is associated with an AUC-ROC significantly greater than 0.50.
To evaluate the effect of unplanned EVD obstruction on the functional outcome assessed on the day of hospital discharge and at 3±1 months. | From EVD insertion to month 3 (± 1 month) after IVH.
  Functional outcome will be considered unfavorable if the modified Rankin scale is 2 or higher, and favorable otherwise. A multivariate analysis involving risk factors for poor functional outcome (dependent variable) and incorporating the occurrence of at least one episode of unplanned EVD obstruction (explanatory variable) will be conducted. If the 95% confidence interval does not include the value 1, then the variable will be retained as an independent risk factor for the occurrence of the dependent variable. As an explanatory variable, we will test, in separate models, the occurrence of at least one episode of unplanned obstruction and the occurrence of at least two episodes.
To evaluate whether the Graeb-EVD, original Graeb, and modified Graeb scores are useful in predicting an EVD-related neuromeningeal infection. | From EVD insertion to ICU discharge up to 6 months.
  Neuromeningeal infection is defined as the administration of antimicrobial therapy for this specific indication for at least 10 days. The predictive performance will be assessed through the area under the receiver operating characteristics curve.
To evaluate the effect of unplanned EVD obstruction on the need for internalization of the ventricular shunt (ventriculoperitoneal or ventriculoatrial shunt). | From EVD insertion to ICU discharge up to 6 months.
  A multivariate analysis involving risk factors for the need for internalization of the ventricular shunt (dependent variable) and incorporating the occurrence of at least one episode of unplanned EVD obstruction (explanatory variable) will be conducted. If the 95% confidence interval does not include the value 1, then the variable will be retained as an independent risk factor for the occurrence of the dependent variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No